CLINICAL TRIAL: NCT03367858
Title: Motivational Interviewing and Neuroimaging With Adolescents
Acronym: MINA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rhode Island (Other)
Responsible Party: Principal Investigator, Sarah Feldstein Ewing, Professor, University of Rhode Island
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5R01AA023658 (NIH)
Record Dates: First submitted 2017-11-29; First posted 2017-12-11 (Actual); Results first posted 2023-11-29 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Alcohol Use, Unspecified
MeSH Terms: conditions — Alcohol Drinking | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motivational Interviewing (MI) (Experimental): This randomly assigned group receives two 60-minute 1:1 sessions of motivational interviewing.
  Interventions: Behavioral: Motivational Interviewing (MI)
- Brief Adolescent Mindfulness (BAM) (Active Comparator): This randomly assigned group receives two 60-minute 1:1 sessions of Brief Adolescent Mindfulness.
  Interventions: Behavioral: Brief Adolescent Mindfulness (BAM)

INTERVENTIONS:
Behavioral: Motivational Interviewing (MI) — Motivational interviewing introduced a conversation about alcohol use, and the personally-experienced consequences of problem drinking. The MI sessions explored youths' stories around their substance use, the factors in youths' lives that support problem drinking (e.g., what they like about drinking), and the consequences of their recent or previous problem drinking (e.g., getting in trouble). Youth were provided personalized feedback about how their problem drinking compared to age-matched norms in the U.S. The ultimate goal of the MI sessions was to engage youth in a thoughtful conversation about their problem drinking with an eye to bolstering and supporting youths' own inherent drive for behavior change.
  Arms: Motivational Interviewing (MI)
Behavioral: Brief Adolescent Mindfulness (BAM) — Brief Adolescent Mindfulness introduced a conversation about what mindfulness is, and ways that it might be personally-relevant to adolescents' current experiences. This manualized treatment introduced concepts of eastern thought in a manner articulated to adolescents. Treatment included a discussion of factors in the youth's life that could be positively impacted by using or engaging mindful approaches (e.g., current experiences of stress) and a link to how mindful approaches might be applicable or relevant to the adolescent's problem drinking. The ultimate goal was to engage youth in a thoughtful conversation about BAM and how eastern thought and mindful approaches could unburden some aspects of their current lived experiences.
  Arms: Brief Adolescent Mindfulness (BAM)

SUMMARY:
This is a randomized controlled trial to examine the impact of two brief interventions on adolescent and young adult alcohol use behaviors and related brain response. The interventions being compared are motivational interviewing (MI) and brief adolescent mindfulness (BAM).

ELIGIBILITY:
Inclusion Criteria:

* within the specified age range
* >= 1 past two month binge drinking episode
* right-handed
* proficient in English
* agree to be contacted for the 3, 6, and 12 month follow ups
* informed consent of a parent/guardian, if under 18 years old
* informed assent/consent of participating youth

Exclusion Criteria:

* > 3 past-month instances of non-nicotine and/or non-cannabis substance use (e.g., methamphetamine)
* evidence of brain injury/illness or neurological disorder including psychosis
* lifetime loss of consciousness >= 2 min
* unremovable metal on/in body, or other functional magnetic resonance imaging (fMRI) contraindications (e.g., pregnancy)

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 204 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2020-01-21 (Actual); Study Completion 2020-01-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Feldstein Ewing, PhD, Principal Investigator — University of Rhode Island
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

REFERENCES:
- [Derived] Dash GF, Chung T, Yang M, Bryan AD, Hudson KA, Feldstein Ewing SW. Examining the influence of adolescent:provider alliance on youth hazardous drinking: Findings from a randomized controlled trial. Addict Behav. 2023 Jan;136:107499. doi: 10.1016/j.addbeh.2022.107499. Epub 2022 Sep 21. PMID 36166981

RESULTS

PARTICIPANT FLOW:
Period: Intervention + Baseline Scan
Arm/Group | Motivational Interviewing (MI) | Brief Adolescent Mindfulness (BAM)
Started | 101 | 103
Completed | 97 | 101
Not Completed | 4 | 2
Not completed — Unable to adhere to session timeline | 2 | 2
Not completed — Withdrawal by Subject | 2 | 0
Period: 3 Month Follow Up
Arm/Group | Motivational Interviewing (MI) | Brief Adolescent Mindfulness (BAM)
Started | 97 (Participants must have completed baseline scan to be eligible for the 3 Month Follow Up scan) | 101 (Participants must have completed baseline scan to be eligible for the 3 Month Follow Up scan)
Completed | 81 | 87
Not Completed | 16 | 14
Not completed — Lost to Follow-up | 8 | 3
Not completed — Moved out of study area | 2 | 6
Not completed — Unable to adhere to session timeline | 1 | 3
Not completed — MRI contraindication | 2 | 1
Not completed — Incarcerated | 0 | 1
Not completed — Withdrawal by Subject | 3 | 0
Period: 6 Month Follow Up
Arm/Group | Motivational Interviewing (MI) | Brief Adolescent Mindfulness (BAM)
Started | 81 (For analysis purposes, only participants with complete scan data (baseline + 3 Month) were followed) | 87 (For analysis purposes, only participants with complete scan data (baseline + 3 Month) were followed)
Completed | 76 | 84
Not Completed | 5 | 3
Not completed — Lost to Follow-up | 5 | 2
Not completed — Withdrawal by Subject | 0 | 1
Period: 12 Month Follow Up
Arm/Group | Motivational Interviewing (MI) | Brief Adolescent Mindfulness (BAM)
Started | 81 (For analysis purposes, only participants with complete scan data (baseline + 3 Month) were followed) | 87 (For analysis purposes, only participants with complete scan data (baseline + 3 Month) were followed)
Completed | 78 | 83
Not Completed | 3 | 4
Not completed — Lost to Follow-up | 3 | 3
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Motivational Interviewing (MI) | Brief Adolescent Mindfulness (BAM) | Total
Number analyzed (Participants) | 101 | 103 | 204
Age, Continuous [Mean (Standard Deviation); unit: years] — Calculated using date of birth and baseline visit date.
  years | 18.83 (1.03) | 18.54 (1.08) | 18.68 (1.06)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 63 | 62 | 125
  Male | 33 | 34 | 67
  Genderqueer / Gender neutral | 4 | 6 | 10
  Transgender | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 13 | 34
  Not Hispanic or Latino | 79 | 89 | 168
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 8 | 12 | 20
  Native Hawaiian or Other Pacific Islander | 2 | 3 | 5
  Black or African American | 2 | 4 | 6
  White | 71 | 64 | 135
  More than one race | 11 | 15 | 26
  Unknown or Not Reported | 5 | 4 | 9
Region of Enrollment [Number; unit: participants]
  United States | 101 | 103 | 204
Alcohol-related Problems [Mean (Standard Deviation); unit: units on a scale] — Rutgers Alcohol Problem Index (RAPI) is a 23 item measure scored on a 5 point Likert scale. Values are sum scores (no reverse coded items). Possible range is 0 - 92, with higher scores indicating greater endorsement of alcohol related problems.
  units on a scale | 8.98 (13.08) | 6.13 (6.60) | 7.54 (10.40)

OUTCOME MEASURES:

1. Primary Outcome: Alcohol-related Problems
Description: Rutgers Alcohol Problems Index (RAPI) to assess alcohol-related problems. Minimum individual value = 0; maximum individual value = 92. Higher scores mean more alcohol-related problems.
Time Frame: assessed at baseline, and 3-, 6-, and 12-month post-treatment follow ups; 12-month follow up reported
Population: Youth with full problem drinking data at all follow up time points were included in treatment outcome analyses.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Motivational Interviewing (MI) | Brief Adolescent Mindfulness (BAM)
Number analyzed (Participants) | 77 | 86
units on a scale | 2.75 (0.45) | 4.88 (0.75)
Statistical Analysis 1: Comparison: Motivational Interviewing (MI) vs Brief Adolescent Mindfulness (BAM); We conducted a repeated measures ANCOVA of Time (Post-Treatment: 3, 6, 12 months) × Treatment (MI, BAM) with the covariate of pre-treatment problem drinking; Test type: Superiority; p = .0173, ANCOVA — At 12 month follow up

ADVERSE EVENTS:
Time Frame: Duration of participant participation (baseline through 12 month follow up).
Arm/Group | Motivational Interviewing (MI) | Brief Adolescent Mindfulness (BAM)
All-Cause Mortality (participants affected / at risk) | 0/101 | 0/103
Serious Adverse Events (participants affected / at risk) | 0/101 | 0/103
Other Adverse Events (participants affected / at risk) | 0/101 | 0/103

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-10-03): https://cdn.clinicaltrials.gov/large-docs/58/NCT03367858/Prot_SAP_000.pdf
  • Informed Consent Form (2018-10-03): https://cdn.clinicaltrials.gov/large-docs/58/NCT03367858/ICF_001.pdf